CLINICAL TRIAL: NCT02334371
Title: MR-PET for Staging and Assessment of Operability in Ovarian Cancer - a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Iris Rutten, Drs., Maastricht University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL50080.068.14
Record Dates: First submitted 2015-01-05; First posted 2015-01-08 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Ovarian Neoplasms
Keywords: Magnetic Resonance Imaging; Positron-Emission Tomography
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MR-PET (Other): Preoperative whole-body MR-PET with 18F-FDG
  Interventions: Radiation: MR-PET

INTERVENTIONS:
Radiation: MR-PET — The MR-PET will be performed with the Biograph mMR system (Siemens Healthcare, Erlangen, Germany). This system integrates a 3Tesla MRI and PET scan which makes simultaneous acquisition of whole-body MRI and PET images possible. The Biograph mMR holds the CE mark and was FDA approved in June 2011. The Biograph mMR is intended to be used in the Academical hospita! Maastricht for standard patient care. The radiotracer that will be used is 18F-Iabeled fluorodeoxyglucose (18F-FDG), according to standard PET -protocol.
  Other Names: MRI-PET; PET-MRI; PET-MR

SUMMARY:
The importance of selecting patients with ovarian cancer who will benefit from either primary debulking surgery or neoadjuvant chemotherapy followed by interval debulking surgery has been acknowledged worldwide but the optimal diagnostic modality to serve in this matter remains to be discovered. We believe that combined magnetic resonance imaging and positron emission tomography (MR-PET) can be of great clinical value in preoperative staging of patients with ovarian cancer.

DETAILED DESCRIPTION:
Recently, the academic hospital Maastricht invested in an integrated MR-PET system (Biograph mMR, Siemens Healthcare, Erlangen, Germany), ready to use for routine clinical application. Applications of this system are numerous and various types of cancer, including ovarian cancer, could benefit from the possibilities. The whole-body MR-PET system integrates the strengths of MRI and PET within a single examination. MRI provides anatomic detail in staging local tumor extent due to its high soft tissue resolution and advanced functional techniques such as DWI further enhance both local and distant lesion detection and characterisation. PET imaging complements this structural and functional information with molecular imaging technology useful in staging of adenopathy and metastatic spread. These characteristics contribute to a wide spectrum of possible clinical oncological applications, from primary tumor detection to local and distant staging, selection of patients for neoadjuvant therapy and assessment of response to chemotherapy and finally evaluation of recurrent disease.

The importance of selecting patients with ovarian cancer who will benefit from either primary debulking surgery or neoadjuvant chemotherapy followed by interval debulking surgery has been acknowledged worldwide but the optimal diagnostic modality to serve in this matter remains to be discovered. We believe that combined magnetic resonance imaging and positron emission tomography (MR-PET) can be of great clinical value in preoperative staging of patients with ovarian cancer. Both positron emission tomography (PET), computed tomography (CT) and magnetic resonance imaging (MRI) have proved to be useful in ovarian cancer staging but understaging due to difficulties in depicting peritoneal dissemination remains a great problem. In conclusion, the best method for staging ovarian cancer and assessing operability remains to be discovered, hence this study.

ELIGIBILITY:
Inclusion Criteria:

* Expected FIGO stage IIB-IV epithelial ovarian carcinoma
* Scheduled for primary debulking or interval debulking surgery
* Written informed consent

Exclusion Criteria:

* Patients estimated to have more benefit from chemotherapy
* Ineligibility to undergo MR-PET examination (Non-MR compatible metallic implants or foreign bodies (ferromagnetic aneurysm clip, pacemaker, neurostimulation system, metal splinters etcetera) or claustrophobia)
* Pregnant or lactating patients.
* Incapacitated subjects

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance | 6 months
  Diagnostic performance of MR-PET compared to CT for characterisation of primary tumour, detection of tumour sites in the peritoneal cavity, retroperitoneum or liver, detection of lymphadenopathy and distant metastases and assessment of tumour stage and operability.

CONTACTS AND LOCATIONS:
Overall Officials: Toon Van Gorp, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qayyum A, Coakley FV, Westphalen AC, Hricak H, Okuno WT, Powell B. Role of CT and MR imaging in predicting optimal cytoreduction of newly diagnosed primary epithelial ovarian cancer. Gynecol Oncol. 2005 Feb;96(2):301-6. doi: 10.1016/j.ygyno.2004.06.054. PMID 15661212
- [Background] Kumar Dhingra V, Kand P, Basu S. Impact of FDG-PET and -PET/CT imaging in the clinical decision-making of ovarian carcinoma: an evidence-based approach. Womens Health (Lond). 2012 Mar;8(2):191-203. doi: 10.2217/whe.11.91. PMID 22375721
- [Background] De Iaco P, Musto A, Orazi L, Zamagni C, Rosati M, Allegri V, Cacciari N, Al-Nahhas A, Rubello D, Venturoli S, Fanti S. FDG-PET/CT in advanced ovarian cancer staging: value and pitfalls in detecting lesions in different abdominal and pelvic quadrants compared with laparoscopy. Eur J Radiol. 2011 Nov;80(2):e98-103. doi: 10.1016/j.ejrad.2010.07.013. Epub 2010 Aug 4. PMID 20688446
- [Background] Wakefield JC, Downey K, Kyriazi S, deSouza NM. New MR techniques in gynecologic cancer. AJR Am J Roentgenol. 2013 Feb;200(2):249-60. doi: 10.2214/AJR.12.8932. PMID 23345344
- [Background] Booth SJ, Turnbull LW, Poole DR, Richmond I. The accurate staging of ovarian cancer using 3T magnetic resonance imaging--a realistic option. BJOG. 2008 Jun;115(7):894-901. doi: 10.1111/j.1471-0528.2008.01716.x. PMID 18485169
- [Background] Fujii S, Matsusue E, Kanasaki Y, Kanamori Y, Nakanishi J, Sugihara S, Kigawa J, Terakawa N, Ogawa T. Detection of peritoneal dissemination in gynecological malignancy: evaluation by diffusion-weighted MR imaging. Eur Radiol. 2008 Jan;18(1):18-23. doi: 10.1007/s00330-007-0732-9. Epub 2007 Aug 14. PMID 17701040
- [Background] Partovi S, Kohan A, Rubbert C, Vercher-Conejero JL, Gaeta C, Yuh R, Zipp L, Herrmann KA, Robbin MR, Lee Z, Muzic RF Jr, Faulhaber P, Ros PR. Clinical oncologic applications of PET/MRI: a new horizon. Am J Nucl Med Mol Imaging. 2014 Mar 20;4(2):202-12. eCollection 2014. PMID 24753986
- [Background] Michielsen K, Vergote I, Op de Beeck K, Amant F, Leunen K, Moerman P, Deroose C, Souverijns G, Dymarkowski S, De Keyzer F, Vandecaveye V. Whole-body MRI with diffusion-weighted sequence for staging of patients with suspected ovarian cancer: a clinical feasibility study in comparison to CT and FDG-PET/CT. Eur Radiol. 2014 Apr;24(4):889-901. doi: 10.1007/s00330-013-3083-8. Epub 2013 Dec 11. PMID 24322510